CLINICAL TRIAL: NCT00802542
Title: In-practice Evaluation of Atacand 16mg Antihypertensive Effect
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Janis Dobelis, AstraZeneca MC Latvia
Other Study IDs: NIS-CLV-ATA-2008/1
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Essential Hypertension
Keywords: Hypertension; blood pressure; Atacand
MeSH Terms: conditions — Essential Hypertension; Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Adult patients with mild or moderate essential hypertension who do not tolerate ACE inhibitors because of cough, already treated with Atacand 8mg for 2-4 weeks, who have not reached the blood pressure treatment goal and the doctor has decided to increase the Atacand dose to 16mg as per SmPC.

SUMMARY:
The purpose of this study is to prove in practice the effectiveness of Atacand 16 mg in reducing blood pressure after 4 weeks of administration and the importance of administration of adequate doses

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with mild (140-159/90-99 mgHg) to moderate (160-179/100-109 mmHg) essential hypertension, already treated with Atacand 8mg for 2-4 weeks, who have not reached the blood pressure treatment goal at least <140/90 mgHg and the doctor has decided
* Signed and dated Patient Informed Consent (ICF)

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients of Atacand.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: out-patient departments
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Decrease in blood pressure | once after 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Agrita Hartmane, Study Director — AstraZeneca
Locations (4):
- Latvia (4):
  - Research site, Daugavpils
  - Research site, Jelgava
  - Research site, Liepāja
  - Research Site, Riga